CLINICAL TRIAL: NCT01487889
Title: Polyunsaturated Fatty Acids in Child Nutrition - A German Multimodal Optimisation Study
Brief Title: Polyunsaturated Fatty Acids in Child Nutrition
Acronym: PINGU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Child Nutrition, Dortmund (Other)
Collaborators: Dr. von Hauner Children's Hospital, Germany (Unknown); University of Potsdam (Other); Pediatric Clinic Dortmund, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PINGU0911DO
Record Dates: First submitted 2011-09-15; First posted 2011-12-08 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Fatty Acid Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rapeseed oil (Experimental): Study group receive commercial vegetable-potato-meat-meals containing rapeseed oil as part of complementary food
  Interventions: Other: Fatty acid composition of complementary food
- Fatty fish (Experimental): Study group receive 2 times per week a vegetable-potato-meat-meals as part of complementary food.
  Interventions: Other: Fatty acid composition of complementary food
- Corn oil (Active Comparator): Study group receive commercial vegetable-potato-meat-meals containing corn oil as part of complementary food
  Interventions: Other: Fatty acid composition of complementary food

INTERVENTIONS:
Other: Fatty acid composition of complementary food — Groups receive commercial vegetable-potato-meat-meals as part of complementary food which differs in the fatty acid composition

SUMMARY:
Primary objective of this study is to examine the effects of 2 different approaches of dietary strategies to optimise fatty acid composition in complementary food on infant's fatty acid status and its consequences on cognitive and visual development.

Subjects are randomly assigned to one of three groups:

* Rapeseed oil (high in n-3 PUFA and small n-6:n-3 ratio to support endogenous n- 3 LC-PUFA metabolism)
* Fatty fish (preformed n-3 LC-PUFA, especially DHA)
* Corn oil (as control group, high in n-6 PUFA, common in complementary food).

The intervention starts with the beginning of complementary feeding as generally recommended between 4 to 6 months of age and ends at the age of 10 months. For this period of time subjects of all groups receive commercial vegetable-potato-meat-meals as part of complementary food which only differs in the fatty acid composition.

DETAILED DESCRIPTION:
A well balanced supply of polyunsaturated fatty acids, in particular the omega-3 long chain docosahexaenoic acid (DHA), in early childhood is essential for children's cognitive and visual development. DHA can either be supplied preformed in the diet (e.g. via fatty fish) or synthesised by conversion of its essential precursor alpha-linolenic acid (e.g. via rapeseed oil). The study examines the effect of two different approaches to optimise infants´ fatty acid status.

The study sample consists of healthy newborns and their mothers (3 x 57 infants according to a priori power calculation) who are enrolled in delivery hospitals in the region of Dortmund, Germany. In total, the individual study program covers the first 10 months of infant's life. Biomarkers of fatty acid status from the mother are collected 8 weeks pp for the estimation of pre- and perinatal fatty acid supply. Additionally, information on maternal diet during pregnancy and after delivery is assessed. The intervention covers the period of complementary feeding (from 4 to 6 months of age until 10 months of age). In all groups the specific study food is given 5 to 7 times a week, whereas 2 of these are fish meals in the fatty fish group. At the age of 4 and 10 months blood samples are collected from the infants to examine the effect on blood fatty acid status. Parameters of visual and cognitive development are also assessed at the age of 4 and 10 months using VEP examinations and Bayley scales. Infants´ dietary intake is assessed from the end of the 2 months until 10 months of age using continuous weighed dietary records.

ELIGIBILITY:
Inclusion Criteria:

* a term healthy newborn infant ( birth weight > 2500 g, gestational age > 37 weeks
* German speaking mother
* the intention of the mother to breast-feed the children and to feed study menus at least 5 times per week beginning in the fifth to seventh month of life.

Exclusion Criteria:

* preterm children
* twins

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Infants´ fatty acid status | 10 months after delivery
  Fatty acids (saturated fatty acids, monounsaturated fatty acids, polyunsaturated fatty acids including long-chain polyunsaturated fatty acids) are measured in percent of total fatty acids in erythrocyte membranes, whole plasma, and cheek cells in order to assess the fatty acid composition.

SECONDARY OUTCOMES:
Infants´ visual development | 10 months after delivery
  Infants´ visual development is assessed using the visual evoked potentials method.
Infants´ cognitive development | 10 months after delivery
  Infants´ cognitive development is assessed using the Bayley II scale.
Infants´ haemogram | 10 months after delivery
Infants´antioxidant status | 10 months after delivery
Infants´ body weight | 10 months after delivery
Infants´ dietary intake | from 2 until 10 months after delivery
Maternal dietary intake | pregnancy and first 2 months post partum
Infant's preference for fish | 10 month after delivery
Infant's preference for new flavour | 10 month after delivery
Parental attitudes about fish and feeding strategies | 10 months after delivery
Mother´s fatty acid status | 2 months after delivery
  Fatty acids (saturated fatty acids, monounsaturated fatty acids, polyunsaturated fatty acids including long-chain polyunsaturated fatty acids) are measured in percent of total fatty acids in erythrocyte membranes, whole plasma, cheek cells, and breast milk in order to assess the fatty acid composition.
Infants´ body length | 10 months after delivery
Infant´s head circumference | 10 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Kersting, Professor, Study Director — Research Institute of Child Nutrition
Locations (1):
- Research Institute of Child Nutrition, Dortmund, Germany

REFERENCES:
- [Derived] Libuda L, Mesch CM, Stimming M, Demmelmair H, Koletzko B, Warschburger P, Blanke K, Reischl E, Kalhoff H, Kersting M. Fatty acid supply with complementary foods and LC-PUFA status in healthy infants: results of a randomised controlled trial. Eur J Nutr. 2016 Jun;55(4):1633-44. doi: 10.1007/s00394-015-0982-2. Epub 2015 Jul 14. PMID 26169870